CLINICAL TRIAL: NCT00724620
Title: Open Multicenter Study of Combination Therapy With Weight-Based PEG-IFN Alfa-2b Plus Ribavirin for Treatment of Mexican naïve Patients With Chronic Hepatitis C Infected With Genotype 1. Impact of the Combination Therapy on Sustained Virological Response and Tolerability, in These Patients.
Brief Title: PEG-IFN Alfa-2b Plus Ribavirin for Treatment of Mexican naïve Patients With Chronic Hepatitis C Infected With Genotype 1 (Study P04511)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04511
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early Responders (ER) (Experimental): All patients will receive peginterferon alfa-2b 1.5 ug/kg administered subcutaneously (SC) once weekly in combination with ribavirin (800-1200 mg/day) administered orally (PO) for a minimum period of 12 weeks. Patients who have responded to therapy at Treatment Week 12 (ie, who are Early Responders defined by HCV-RNA[-] at Treatment Week 12) will continue the combined treatment for a total of 48 weeks and will complete 24 weeks of follow up to determine the Sustained Viral Response (SVR).
  Interventions: Biological: Peginterferon alfa-2b (SCH 054031); Drug: Ribavirin (SCH 018908)
- Slow Responders (SR): Decrease in viral load >=2 log (Experimental): All patients will receive peginterferon alfa-2b 1.5 ug/kg administered subcutaneously (SC) once weekly in combination with ribavirin (800-1200 mg/day) administered orally (PO) for a minimum period of 12 weeks. Patients who have a slow response to therapy at Treatment Week 12 (ie, Slow Responders who are not HCV-RNA[-] at Treatment Week 12 but decrease >=2 log) will continue the combined treatment for a total of 72 weeks and will complete 24 weeks of follow up to determine the Sustained Viral Response (SVR).
  Interventions: Biological: Peginterferon alfa-2b (SCH 054031); Drug: Ribavirin (SCH 018908)
- Nonresponders (NR): Decrease in viral load <2 log (Experimental): All patients will receive peginterferon alfa-2b 1.5 ug/kg administered subcutaneously (SC) once weekly in combination with ribavirin (800-1200 mg/day) administered orally (PO) for a minimum period of 12 weeks. Patients who have not responded to therapy at Treatment Week 12 (ie, Nonresponders who are not HCV-RNA[-] at Week 12 of Treatment and/or have a decrease in viral load <2 log) will stop treatment at Treatment Week 12.
  Interventions: Biological: Peginterferon alfa-2b (SCH 054031); Drug: Ribavirin (SCH 018908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 054031) — All patients will receive peginterferon alfa-2b 1.5 ug/kg administered subcutaneously (SC) once weekly in combination with ribavirin (800-1200 mg/day) administered orally (PO) for a minimum period of 12 weeks. The total treatment duration will be as follows: 48 weeks for Early Responders, 72 weeks for Slow Responders, and 12 weeks for Nonresponders.
  Other Names: PegIntron
Drug: Ribavirin (SCH 018908) — All patients will receive peginterferon alfa-2b 1.5 ug/kg administered subcutaneously (SC) once weekly in combination with ribavirin (800-1200 mg/day) administered orally (PO) for a minimum period of 12 weeks. The total treatment duration will be as follows: 48 weeks for Early Responders, 72 weeks for Slow Responders, and 12 weeks for Nonresponders.
  Other Names: Rebetol

SUMMARY:
This study aims to evaluate the efficacy and safety of peginterferon alfa-2b plus weight-based ribavirin as initial treatment in chronic hepatitis C virus (HCV) genotype 1 patients. All patients will receive peginterferon alfa-2b plus oral ribavirin for 12 weeks. At the end of this period, quantitative PCR will be used to determine the Early Viral Response (EVR) at this point of treatment. Total treatment duration will be 48 weeks for Early Responders, 72 weeks for Slow Responders, and 12 weeks for Nonresponders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had given their informed consent in writing.
* Adult patients, older than 18 and younger than 65 years.
* Be hepatitis C treatment-naïve patients.
* Patients should have been assessed at entry and their METAVIR score of fibrosis determined as F2, F3 or F4.
* Patients should have been diagnosed, at treatment week 0, visit 1 (V1), chronic hepatitis C determined through a positive HCV-RNA test by RT-PCR (reverse transcriptase-polymerase chain reaction) assay.
* Patients with F4 METAVIR score should have a Class A score in Child-Pugh classification, in which the following criteria should be met: Prothrombin time <=3.0 seconds; Absence of ascites; Absence of encephalopathy.
* Patients should have a compensated liver disease meeting the following minimum hematologic, biochemical and serologic criteria: Hemoglobin: >=12 g/dL in women and >=13 g/dL in men; Leukocyte count: >=3 000/mm^3; Neutrophil count: >=1 500/mm^3; Platelet count: >=80 000/mm^3; Direct bilirubin, albumin, serum creatinine: within normal ranges.
* Patients with a history of addiction should have abstained from consuming drugs for at least two years. All patients must be willing not to consume alcohol during the study.
* The investigator should confirm that sexually active women in child-bearing age are using adequate contraceptive methods.
* Neither the participating women nor the partners of participating men shall get pregnant during the study.
* Women must not get pregnant or be breast-feeding during the study period.

Exclusion Criteria:

* Having participated in any other clinical study within 30 days prior to visit at week 0 (V1) of this study treatment.
* Suffering from another liver disease other than chronic hepatitis C, such as: Hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, Autoimmune hepatitis , Alcoholic liver disease, Obesity-induced liver disease, Drug-induced liver disease.
* With a known coinfection with HIV or HBV.
* With evidence of decompensated liver diseases, such as history or presence of ascites, jaundice, bleeding varices, esophageal or gastric varices or hepatic encephalopathy.
* With a history of hepatocellular carcinoma (HCC).
* With any pre-existing medical condition that may interfere with patient's participation in and/or conclusion of the study, such as: Clinically significant retinal anomalies, Central nervous system (CNS) trauma or convulsive disorders, Poorly controlled diabetes mellitus, Autoimmune diseases (eg, inflammatory intestinal diseases [Crohn's disease, ulcerative colitis], rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis, or symptomatic thyroid disorders), Chronic pneumopathies (eg, chronic obstructive pulmonary disease), Cardiovascular dysfunction or clinically significant electrocardiographic alterations within six months prior to visit at week 0 (eg, angina pectoris, congestive heart failure, recent heart attack, severe hypertension or significant arrhythmia), Suspected hypersensitivity to any interferon or to Ribavirin, Any organ transplantation, except corneal and hair transplantation
* With signs of suspected or active cancer or history of cancer within past five years (except for basocellular skin carcinomas receiving adequate treatment)
* With addiction, such as alcoholism (>=40 g/day), intravenous (IV) drugs and inhaled drugs. Patients who have received methadone, buprenorphine hydrochloride or butorphanol tartrate within past two years may not be admitted either.
* Suffering from any other condition that, in the investigator's opinion, would either make the patient inadequate for admission to study or affect his/her participation in and the conclusion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall SVR of chronic hepatitis C Genotype 1 Naïve Mexican patients with different durations of treatment. | SVR will be determined after 48 weeks of treatment and 24 weeks of follow-up in the Early Responders and after 72 weeks of treatment and 24 weeks of follow-up in the Slow Responders.